CLINICAL TRIAL: NCT04653571
Title: Defining the Initial Clinical Symptoms and Characterizing Those Leading to the Discovery of CASPR2
Brief Title: CASPR2 Encephalitis Initial Symptoms
Acronym: iniCASPR2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0760
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: CASPR2-Antibody; Encephalitis Autoimmune; Paraneoplastic Syndromes
Keywords: antibody ; auto-immune encephalitis ; paraneoplastic syndrome ; CASPR2
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Paraneoplastic Syndromes; Cortical Dysplasia-Focal Epilepsy Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CASPR2 encephalitis: Cohort of patients with a CASPR2 antibody-associated auto-immune encephalitis.
  Interventions: Other: CASPR2 encephalitis

INTERVENTIONS:
Other: CASPR2 encephalitis — Defining the initial clinical symptoms and those leading to the diagnosis of CASPR2 antibody associated encephalitis. For that, we will investigate the initial cognitive status, the initial neuropsychological investigations the clinical presentation of the first seizures, and the prodromes assessed by patients at the beginning of their disease. We will also look at the initial EEG records, in order to acknowledge whether the initial cognitive symptoms may be due to unseen seizures.

SUMMARY:
Auto-immune encephalitides involve auto-antibodies targeting the central nervous system, and particularly the synapse and its structure, such as protein CASPR2.

CASPR2 antibody-associated auto-immune encephalitides lead to an inflammation of the limbic system and generate focal temporal seizures and cognitive impairment. Most patients are initially hospitalized because of the temporal seizures (Joubert et al., JAMA Neurology 2016). However, many already show at that time cognitive impairment, which has failed to elicit the appropriate investigations, therefore delaying the diagnosis.

The study will hence investigate precisely the initial, sometimes neglected, clinical symptoms and those leading to the diagnosis, in the cohort of patients suffering from a CASPR2 antibody-associated encephalitis, from the French reference center on paraneoplastic neurological diseases and autoimmune encephalitis.

This way, the study aims to delineate the symptoms that should trigger suspicions of a CASPR2 antibody-associated encephalitis

ELIGIBILITY:
Inclusion Criteria:

* Positive CASPR2-Ab in serum and/or CSF tested by immunohistochemistry on mouse brain slices and confirmed by cell-based assay (CBA) of HEK293 cells expressing CASPR2.
* Diagnosis and follow-up in France
* From 18 to unlimited age

Exclusion Criteria:

* Patients CASPR2-IgG negative in serum and CSF
* Foreign follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a CASPR2 antibody-associated auto-immune encephalitis
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Initial cognitive impairment or clinical presentation of first epileptic seizures. | 8 months
  The retained information will depend on the very first declared symptom: if the patient first showed focal seizures, we will precise the clinical presentation of this seizure. On the other hand, if the patient first showed cognitive symptoms, we will best define this impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme HONNORAT, Pr, Principal Investigator — Service de neuro-oncologie, Hôpital neurologique
Locations (1):
- Service de Neuro-Oncologie, Hôpital Neurologique Pierre Wertheimer, Bron, France

IPD SHARING:
Plan to Share IPD: No